CLINICAL TRIAL: NCT03400358
Title: Uterocervical Angle in the Termination of Second Trimester Pregnancy in Multiparous Women
Brief Title: Uterocervical Angle in the Pregnancy Termination of Multiparous Women
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2016/12.5
Record Dates: First submitted 2018-01-06; First posted 2018-01-17 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Medical; Abortion, Fetus; Second Trimester Abortion
Keywords: uterocervical angle; multiparous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical abortion: 150 singleton multiparous patients are planning to complete the study period. Study group constitute of second trimester pregnancies between 14-24 weeks of gestation. All participants were multiparous and had no systemic illnesses. The uterocervical angle will be measured in all participants before the induction of labor.
  Interventions: Other: uterocervical angle

INTERVENTIONS:
Other: uterocervical angle — the angle between cervical canal and anterior uterine wall is measured sonographically.

SUMMARY:
To evaluate the uterocervical angle (UCA) in the prediction of second trimester termination success of multiparous women.

DETAILED DESCRIPTION:
Medical termination of pregnancy is a common procedure in obstetrics. In recent years, uterocervical angle (UCA) emerged as a new ultrasound parameter in the prediction of labor. Dziadosz et al concluded that the performance of UCA was even better than the cervical length in their cohort. A wide UCA during second trimester shown to have an increased risk of preterm labor and narrow angle was less likely to have labor.

The investigators are aimed to investigate predictive role of both cervical length and UCA in the termination of second trimester pregnancy.The investigators focused on multiparous women who are taking Foley baloon for the cervical preparation and aim to measure their UCA.

ELIGIBILITY:
Inclusion Criteria:

* multiparous singleton pregnancy
* no previous systemic illnesses

Exclusion Criteria:

* abnormal Pap smear
* history of dilatation and curettage (D&C)
* history of LEEP and cervical conization

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Multiparous pregnant women undergoing medical abortion in the second trimester
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
uterocervical angle | 1 week
  the angle between the cervical canal and anterior uterine wall

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28055026